CLINICAL TRIAL: NCT07159373
Title: Safety and Efficacy Trial of Mass Drug Administration With Moxidectin Versus Ivermectin in Combination With Diethylcarbamazine and Albendazole for Lymphatic Filariasis, Scabies, and Strongyloidiasis in Fiji
Brief Title: Better Options for Lymphatic Filariasis Treatment
Acronym: BOLT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medicines Development for Global Health (Other)
Collaborators: Murdoch Childrens Research Institute (Other); Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDGH-MOX-3003
Record Dates: First submitted 2025-08-26; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Lymphatic Filariasis; Scabies; Strongyloidiasis
Keywords: Moxidectin; Ivermectin; Mass drug administration; Lymphatic filariasis; Scabies; Strongyloidiasis; Cluster-randomized; Diethylcarbamazine; Albendazole
MeSH Terms: conditions — Elephantiasis, Filarial; Scabies; Strongyloidiasis | interventions — Albendazole

STUDY DESIGN:
Intervention Model Description: Open label trial of mass drug administration with two treatment arms cluster-randomized 1:1 by village and stratified by island.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MoxDA (Experimental): Moxidectin + diethylcarbamazine + albendazole
  Interventions: Drug: MoxDA - Moxidectin + Diethylcarbamzine (DEC) + Albendazole
- IDA (Active Comparator): Ivermectin + diethylcarbamazine + albendazole
  Interventions: Drug: IDA - Ivermectin + DEC + albendazole

INTERVENTIONS:
Drug: MoxDA - Moxidectin + Diethylcarbamzine (DEC) + Albendazole — Mass drug administration with moxidectin co-administered with DEC and albendazole (MoxDA).
  Participants who are ineligible to receive moxidectin will be offered modified treatment options:
  1. Children aged ≥ 2 years but < 4 years - DEC, albendazole, and permethrin 5% cream
  2. Participants who have a severe illness, a known or suspected allergy to ivermectin, moxidectin, DEC or albendazole, are pregnant or breastfeeding a baby up to 7 days of age, or are under 2 years of age - permethrin 5% cream (unless allergic)
  Arms: MoxDA
Drug: IDA - Ivermectin + DEC + albendazole — Mass drug administration with ivermectin co-administered with DEC and albendazole (IDA).
  Participants who are ineligible to receive moxidectin will be offered modified treatment options:
  1. Children aged < 2 years or weight < 15 kg - DEC, albendazole, and permethrin 5% cream
  2. Participants who have a severe illness, a known or suspected allergy to ivermectin, moxidectin, DEC or albendazole, are pregnant or breastfeeding a baby up to 7 days of age, or are under 2 years of age - permethrin 5% cream (unless allergic)
  Arms: IDA

SUMMARY:
The goal of this clinical trial is to learn if mass drug administration with moxidectin in combination with diethylcarbamazine, and albendazole (MoxDA) can treat lymphatic filariasis, scabies and strongyloidiasis in children and adults living in communities where these diseases are common. The main questions it aims to answer are:

1. Does MoxDA clear infection in people with lymphatic filariasis ?
2. Does MoxDA cause any medical problems in infected and uninfected people?

Researchers will compare MoxDA with ivermectin given together with diethylcarbamazine and albendazole (IDA) to see if it works better to clear infection and does not cause any more medical problems.

Participants will:

1. Be tested to see if they are infected with the parasites that cause lymphatic filariasis, scabies and strongyloidiasis
2. Take 3 single doses of MoxDA or IDA, 12 months apart
3. Visit their village centre once or twice in the 1 week after each treatment for safety checkups

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent.
2. Resident in one of the study locations.

Exclusion Criteria:

There are no exclusion criteria to participation in the study.

Treatment Exclusion Criteria:

Participants are ineligible to receive the treatment regimen allocated to their village if they meet any of the following criteria:

1. Severe illness (any illness that is severe enough to interfere with activities of daily living);
2. Known or suspected allergy to ivermectin, moxidectin, diethylcarbamazine or albendazole;
3. Pregnant;
4. Breastfeeding a baby within 7 days of birth;
5. Age < 4 years for villages randomised to moxidectin, diethylcarbamazine, and albendazole (MoxDA); or
6. Age < 2 years or weight < 15 kg for villages randomized to ivermectin, diethylcarbamazine and albendazole (IDA).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of microfilariae (Mf)-positive participants at Baseline who are Mf-negative at Month 12 following treatment with MoxDA or IDA | 12 months post-treatment
  Lymphatic filariasis (LF) Mf measured by ultrafiltration
Incidence and severity of adverse events | 7 days, 12 months and 24 months post-treatment
  Frequency, type, and severity of adverse events reported by treatment group

SECONDARY OUTCOMES:
Proportion of Mf-positive participants at Baseline who are Mf-negative at Month 24 following treatment with MoxDA or IDA | 24 months post-treatment
  LF Mf measured using ultrafiltration
Mean Mf density and mean change from Baseline at Months 12 and 24 following treatment with MoxDA or IDA in participants who are Mf-positive at Baseline | 12 and 24 months post-treatment
  LF Mf measured using ultrafiltration
Proportion of participants who are circulating filarial antigen (CFA)-positive at baseline who become CFA-negative at Months 12 and/or 24 following treatment with MoxDA or IDA | 12 and 24 months post-treatment
  CFA measured using rapid lateral flow assay
Change in community prevalence of LF, as measured by Mf, at Months 12 and 24 following annual MDA with MoxDA or IDA, in addition to directed treatment of individuals who are Mf positive at 3-monthly assessments between Months 12 and 24 | 12 and 24 months post-treatment
  LF Mf measured using ultrafiltration
Change in community prevalence of LF, as measured by CFA, at Months 12 and 24 following annual MDA with MoxDA or IDA, in addition to directed treatment of individuals who are Mf positive at 3-monthl | 12 and 24 months post-treatment
  CFA measured using rapid lateral flow assay
Proportion of participants with presence of Mf between Month 12 and Month 24 among those who were Mf positive at Month 12 following treatment with MoxDA or IDA | 12 to 24 months post-treatment
  LF Mf measured using ultrafiltration
Time to first detection of Mf in participants with presence of Mf between Month 12 and Month 24 among those who were Mf positive at Month 12 following treatment with MoxDA or IDA | 12 to 24 months post-treatment
  Lf Mf measured using ultrafiltration
Community acceptability of MDA with MoxDA or IDA assessed by surveys, focus group discussions, and/or key informant interviews before Baseline and approximately 2 months following MDA at Baseline and Month 12 | Pre- and post-treatment at Baseline and post-treatment at Month 12
Change in community prevalence of scabies and impetigo at Months 12 and 24 following annual community MDA with MoxDA or IDA, in addition to directed treatment of individuals who are Mf positive at 3-monthly assessment between Months 12 and 24 | 12 and 24 months post-treatment
  Scabies and impetigo measured using modified International Alliance for the Control of Scabies (IACS) criteria based on examination of normally exposed skin
Change in community seroprevalence of S. stercoralis at Months 12 and 24 following annual MDA with MoxDA or IDA, in addition to directed treatment of individuals who are Mf positive at 3-monthly assessments between Months 12 and 24 | 12 and 24 months post-treatment
Change in community prevalence of LF, as measured by Mf and CFA, at Months 12 and 24 following annual MDA with MoxDA or IDA, in addition to directed treatment of individuals who are Mf positive at 3-monthly assessments between Months 12 and 24 | 12 and 24 months post-treatment
  LF Mf measured using ultrafiltration and CFA measured using rapid lateral flow assay

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health and Medical Services Fiji, Suva, Fiji

IPD SHARING:
Plan to Share IPD: Undecided